CLINICAL TRIAL: NCT05321836
Title: EFFECTS OF COMBINED GLUCOSAMINE/CHONDROITIN WITH STRUCTURED PHYSICAL THERAPY PROGRAM ON KNEE OSTEOARTHRITIS: A RANDOMIZED CONTROL TRAIL
Brief Title: GLUCOSAMINE/CHONDROITIN and PHYSICAL THERAPY EFFECTS ON OLDER POPULATION WITH KNEE OSTEOARTHRITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad salman, PT (Other)
Responsible Party: Sponsor-Investigator, Muhammad salman, PT, Principal researcher, Neuro Counsel Hospital, Pakistan
Organization: Neuro Counsel Hospital, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 333
Record Dates: First submitted 2022-03-26; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: OA, Chondratin sulfate, glucosamine, Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: two groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): chondritin sulfate 1500/1200mg
  Interventions: Other: Glucosamine Chondroitin
- experimental group (Experimental): chondritin sulfate plus physiotherapy
  Interventions: Combination Product: glucosamine chondritin & Physiotherapy

INTERVENTIONS:
Other: Glucosamine Chondroitin — control group
  Arms: control group
Combination Product: glucosamine chondritin & Physiotherapy — experimental group
  Arms: experimental group

SUMMARY:
to see the effect of glucosamine chondratin sulfate with and without physiotherapy in knee osteoarthritis

DETAILED DESCRIPTION:
it is a randomized control trail to evaluate the effectiveness of glucosamine chondratin sulfate alone and in combination with physiotherapy on knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years with radiographic evidence of mild to moderate knee OA (Kellgren Lawrence grade II & III 20) who met the ACR clinical 21,
* radiographic classification criteria or confirmation of mild to moderate radiographic evidence of knee OA from a personal physician
* not currently participating in another intervention study

Exclusion Criteria:

* dementia (Mini-Mental State Examination [MMSE]< 24)
* active cancer other than skin cancer
* anemia (participants with an hematocrit (HCT)< 32 (or a hemoglobin below10) were excluded due to possible inability to adequately exercise or the increased potential for increased risk for serious adverse cardiovascular events)
* severe renal insufficiency (serum creat> 2)
* hepatic disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
WOMAC | 6 months
  higher score means worst patient condition and lower score means better

SECONDARY OUTCOMES:
SF-36 | 6 months
  higher score means better patient condition and lower score means worst

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD UMAR, Principal Investigator — the physiotherapy clinic
Locations (1):
- Muhammad Umar, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No